CLINICAL TRIAL: NCT05349188
Title: Re-engineering Precision Therapeutics Through N-of-1 Trials: Feasibility Study of Personalized Trials to Improve Sleep Quality
Brief Title: Feasibility Study of Personalized Trials to Improve Sleep Quality
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Library of Medicine (NLM) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-0239; R01LM012836 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disturbance
Keywords: Sleep; Personalized; N-of-1; Virtual; Feasibility; Melatonin; Sleep Quality
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The study utilizes a multiple crossover design to conduct N-of-1 trials in individuals.
Who Masked: Participant
Masking Description: Participants are blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Melatonin 3 mg (Experimental): Individuals will receive a kit with medication adherence devices containing melatonin 3 mg in one of three smart electronic pill bottles labeled "A," "B," and "C." Participants will not be aware which of the pill bottles contains the 3mg of melatonin. Participants will be randomized to take pills in 6 alternating intervention periods 2 weeks in length. During periods where participants were randomized to receive melatonin 3 mg, they will receive a nightly text notification 1 hour before bed instructing them to take a pill from the corresponding smart pill bottle. The melatonin 3 mg intervention will be administered in 2 intervention periods each 2 weeks in length (4 weeks total).
  Interventions: Dietary Supplement: Melatonin 3 mg
- Melatonin 0.5 mg (Active Comparator): Individuals will receive a kit with medication adherence devices containing melatonin 0.5 mg in one of three smart electronic pill bottles labeled "A," "B," and "C." Participants will not be aware which of the pill bottles contains the 0.5 mg of melatonin. Participants will be randomized to take pills in 6 alternating intervention periods 2 weeks in length. During periods where participants were randomized to receive melatonin 0.5 mg, they will receive a nightly text notification 1 hour before bed instructing them to take a pill from the corresponding smart pill bottle. The melatonin 0.5 mg intervention will be administered in 2 intervention periods each 2 weeks in length (4 weeks total).
  Interventions: Dietary Supplement: Melatonin 0.5 mg
- Placebo Pill (Placebo Comparator): Individuals will receive a kit with medication adherence devices containing the placebo pills in one of three smart electronic pill bottles labeled "A," "B," and "C." Participants will not be aware which of the pill bottles contains the placebo. Participants will be randomized to take pills in 6 alternating intervention periods 2 weeks in length. During periods where participants were randomized to receive the placebo, they will receive a nightly text notification 1 hour before bed instructing them to take a pill from the corresponding smart pill bottle. The placebo will be administered in 2 intervention periods each 2 weeks in length (4 weeks total).
  Interventions: Other: Cellulose placebo pill

INTERVENTIONS:
Dietary Supplement: Melatonin 3 mg — Participants will be provided with a smart pill bottle containing a 4-week supply of 3 mg melatonin pills.
  Arms: Melatonin 3 mg
Dietary Supplement: Melatonin 0.5 mg — Participants will be provided with a smart pill bottle containing a 4-week supply of 0.5 mg melatonin pills.
  Arms: Melatonin 0.5 mg
Other: Cellulose placebo pill — Participants will be provided with a smart pill bottle containing a 4-week supply of cellulose placebo pills.
  Arms: Placebo Pill

SUMMARY:
The purpose of this pilot study is to assess the feasibility of using N-of-1 methods in a virtual research study of melatonin intervention for poor sleep quality. Participants (N=60) will be sent a Fitbit device and 3 smart pill bottles, with one containing 3 mg of melatonin, one containing 0.5 mg of melatonin, and the final bottle containing a placebo pill. The first two weeks will be a baseline period, where no supplement is assigned, but data are collected, including self-report of sleep quality and duration and accelerometer-derived sleep and activity data. After successful completion of the baseline period, participants will be randomized to six 2-week intervention blocks of a 3 mg dose melatonin, a 0.5 mg dose melatonin, and a placebo. At the end of the trial, participants will be asked to complete the System Usability Scale, a satisfaction survey (electronic or phone/video call if they are non-responders), and participate in a virtual interview (such as over Microsoft Teams or a phone call) to inform feasibility and acceptability of protocol requirements, study materials, and personalized reports.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the feasibility of using N-of-1 methods in a virtual research study; to remotely recruit and enroll participants; to assess the feasibility of using a placebo and to determine the feasibility of the proposed methods used to collect and assess participant adherence and response to a wellness strategy (in this case, melatonin for poor sleep quality). This pilot will help determine if an N-of-1 study design, or what has been termed 'Personalized Trials', can have widespread use in future research and clinical practice to address high public health burdens with a high heterogeneity of response. This pilot study will assess feasibility using a Personalized Trials model to evaluate an individual participant's experience with a wellness strategy for self-reported poor sleep quality. Participants (N=60) will be sent a Fitbit device and 3 smart pill bottles, with one containing 3 mg of melatonin, one containing 0.5 mg of melatonin, and the final bottle containing placebo pills. Participants will be asked several questions a day sent via text message about their sleep quality, as well as their stress, fatigue, concentration, confidence, mood, and pain levels to demonstrate relevant secondary impacts of sleep quality. Participants will also have access to several videos explaining the protocol. The study will take place over the course of 14 weeks. The first two weeks will be a baseline period, where no supplement is assigned, but data are collected, including self-report of sleep quality and duration and accelerometer-derived sleep and activity data. After successful completion of the baseline period, participants will be randomized to six 2-week intervention blocks of a 3 mg dose melatonin, a 0.5 mg dose melatonin, and a placebo. At the end of the 14 weeks, a report containing the individual's observed data will be prepared for each participant and electronically sent to them along with a satisfaction survey (electronic, or phone/video call if they are non-responders).

After the end of the 14-week trial, participants will receive a summary of their observed data in a personalized report. Creating this type of report will help to assess the feasibility of using a N-of-1 trial design through user-acceptability of sleep quality and wellness-related data visualizations, and the ability to choose preferred intervention (if any) based on the data. Participants will be asked to complete the System Usability Scale, a satisfaction survey (electronic or phone/video call if they are non-responders), and participate in a virtual interview (such as over Microsoft Teams or a phone call) to inform feasibility and acceptability of protocol requirements, study materials, and personalized reports.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Fluent in English
* Ability to take melatonin and a placebo
* Self-report of disrupted sleep symptoms using the Insomnia Symptom Questionnaire (ISQ)
* Owns and can regularly access a smartphone capable of receiving text messages
* Owns and can regularly access an e-mail account
* Lives in the United States
* Agreement to adhere to lifestyle considerations including wearing a Fitbit device day and night and potentially adapting their current melatonin routine to fit the protocol throughout study duration

Exclusion Criteria:

* Age < 18 years old
* Women who are pregnant or breastfeeding
* Individuals diagnosed with depression, seasonal affective disorder, schizophrenia, autoimmune disease, or asthma
* Individuals taking MAO inhibitors or corticosteroids
* Individuals diagnosed with low blood pressure
* Clinical diagnosis of a sleep disorder (e.g., Narcolepsy, Circadian Rhythm Sleep-Wake Disorders, Periodic Limb Movement Disorder, Restless Leg Syndrome, Obstructive Sleep Apnea etc.)
* Deemed unable to complete the study protocol as a result of cognitive impairment, severe medical or mental illness, or active or prior substance abuse
* Participation in shift work (evening/night shifts, early morning shifts, rotating shifts, etc.)
* Pilot or flight attendant with frequent travel across time zones
* Receiving specialty mental health care for insomnia (e.g., cognitive behavioral therapy for insomnia, medications for insomnia)
* Has even been told by a doctor or healthcare provider that it is not safe to take melatonin
* Does not own or cannot regularly access a smartphone capable of receiving text messages
* Does not possess or cannot regularly access an email account
* Lives outside the United States
* Planned surgeries within 6 months from study start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary.
  Supporting Information: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
  Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

REFERENCES:
- [Derived] Butler M, D'Angelo S, Perrin A, Rodillas J, Miller D, Arader L, Chandereng T, Cheung YK, Shechter A, Davidson KW. A Series of Remote Melatonin Supplement Interventions for Poor Sleep: Protocol for a Feasibility Pilot Study for a Series of Personalized (N-of-1) Trials. JMIR Res Protoc. 2023 Aug 3;12:e45313. doi: 10.2196/45313. PMID 37535419

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Personalized Trial: Participants in Group 1 received all three arms of the study in two-week blocks in the following order: 3 mg melatonin, .5 mg melatonin, placebo, placebo, .5 mg melatonin, 3 mg melatonin.
- Group 2 Personalized Trial: Participants in Group 2 received all three arms of the study in two-week blocks in the following order: placebo, .5 mg melatonin, 3 mg melatonin, 3 mg melatonin, .5 mg melatonin, placebo.
Period: Overall Study
Arm/Group | Group 1 Personalized Trial | Group 2 Personalized Trial
Started | 30 | 30
First Intervention Block (2 Weeks) | 30 | 30
Second Intervention Block (2 Weeks) | 30 | 30
Third Intervention Block (2 Weeks) | 29 | 30
Fourth Intervention Block (2 Weeks) | 29 | 30
Fifth Intervention Block (2 Weeks) | 29 | 30
Sixth Intervention Block (2 Weeks) | 29 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants offered primary outcome
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Personalized Trial | Group 2 Personalized Trial | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (13.1) | 39.4 (12.3) | 41.1 (12.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 11 | 16 | 27
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 16 | 18 | 34
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean System Usability Score (SUS)
Description: The SUS is a validated 10-item questionnaire that asks users to score each item on a Likert scale from Strongly Disagree (rating of 1) to Strongly Agree (rating of 5). The SUS will be presented to the participant as addressing the ease of use, complexity, consistency of the Personalized Trials system as a whole, from recruitment to receipt of the report. Individual results are calculated to arrive at a composite measure out of 100. Participant SUS scores will be averaged together and an overall mean will be reported with standard deviation. Higher scored values correlate to a more usable system, and therefore a better outcome.
Time Frame: Assessed once after the results report has been sent to the participant after completion of the trial (14 weeks from baseline).
Population: Pre-specified to report results at the whole sample level. Though the study utilizes two groups with two treatment orders, this is done to counter-balance the presentation of treatments (3 mg melatonin, .5 mg melatonin, and placebo). Of the 60 participants enrolled in the trial, all were sent the SUS to evaluate the feasibility and acceptability of the trial. Completed survey measures were received for 57 of the 60 (95.0%) participants who were offered the outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Participants in both treatment order groups are combined for analyses of primary and secondary outcomes.
Arm/Group | All Participants
Number analyzed (Participants) | 57
score on a scale | 76.27 (17.09)

2. Primary Outcome: Participant Satisfaction With Personalized Trial Components
Description: Participants will rate their satisfaction with the Personalized N-of-1 Trial overall and with individual elements of the trial in a satisfaction survey administered following the baseline and intervention periods (14 weeks). Means and standard deviations will be reported for each element of satisfaction. Participants will rate their satisfaction on a scale of 1 to 5, with higher scores indicating greater levels of satisfaction.
Time Frame: as for outcome 1
Population: Pre-specified to report results at the whole sample level. Though the study utilizes two groups with two treatment orders, this is done to counter-balance the presentation of treatments (3 mg melatonin, .5 mg melatonin, and placebo). Of the 60 participants enrolled in the trial, all were sent a satisfaction survey to evaluate the feasibility and acceptability of the trial. Completed survey measures were received for 57 of the 60 (95.0%) participants who were offered the outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Pre-specified to report results at the whole sample level. Participants in both treatment order groups are combined for analyses of primary and secondary outcomes.
Arm/Group | All Participants
Number analyzed (Participants) | 57
score on a scale
  "Your Personalized Trial to Improve Sleep Quality." | 4.04 (1.19)
  "Video explanations and demonstrations of study devices and procedures." | 4.40 (.75)
  "Text messaging for reminders." | 3.67 (1.42)
  "Text messaging for survey questions." | 3.47 (1.48)
  "Use of the Fitbit to track your activity and sleep." | 4.58 (.94)
  "Presentation of your results." | 4.51 (.89)

3. Secondary Outcome: Within-Participant Difference in Fitbit Device-Recorded Sleep Duration.
Description: Nightly sleep duration will be assessed by a Fitbit wearable device. Sleep duration will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Sleep duration values over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Nightly sleep duration will be assessed consistently via Fitbit device during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Population: Of the 60 enrolled participants, 55 (91.7%) participants had sufficient Fitbit data to include in analyses.
Measure: Mean (Standard Deviation); unit: minutes per night
Groups:
- Baseline Assessment Period: At the beginning of the study, individuals will undergo two weeks of a baseline assessment period, where no supplement is assigned, but data are collected, including self-report of sleep quality and duration and accelerometer-derived sleep and activity data.
Arm/Group | Baseline Assessment Period | Melatonin 3 mg | Melatonin 0.5 mg | Placebo Pill
Number analyzed (Participants) | 55 | 55 | 55 | 55
minutes per night | 399 (53) | 402 (61) | 398 (54) | 398 (59)

4. Secondary Outcome: Mean Within-Subject Difference in Self-Reported Sleep Quality.
Description: Participants will rate their sleep disturbance using a modified version of the Consensus Sleep Diary administered daily during baseline and intervention periods (14 weeks). Participants will be asked to rate their sleep on a 5-point scale rated from "very poor" to "very good". Levels of daily sleep quality will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period, with higher scores indicating better sleep quality. Changes in sleep quality over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Daily sleep quality will be assessed daily via survey during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each).
Population: Of the 60 enrolled participants, 55 (91.7%) participants had sufficient sleep quality data during the baseline assessment, melatonin .5 mg, and placebo periods, and 54 (90.0%) participants had sufficient sleep quality data during the melatonin 3 mg period to include in analyses.
Measure: Mean (Standard Deviation); unit: score on a scale per day
Arm/Group | Baseline Assessment Period | Melatonin 3 mg | Melatonin 0.5 mg | Placebo Pill
Number analyzed (Participants) | 55 | 54 | 55 | 55
score on a scale per day | 3.13 (.64) | 3.35 (.56) | 3.44 (.55) | 3.38 (.53)

5. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Fatigue.
Description: Fatigue will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0(low) to 10(high). Levels of EMA fatigue will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA fatigue over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA fatigue will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Population: Of the 60 enrolled participants, 55 (91.7%) participants had sufficient EMA data during the baseline assessment, melatonin .5 mg, and placebo periods, and 54 (90.0%) participants had sufficient EMA data during the melatonin 3 mg period to include in analyses.
Measure: Mean (Standard Deviation); unit: units on a scale per period
Arm/Group | Baseline Assessment Period | Melatonin 3 mg | Melatonin 0.5 mg | Placebo Pill
Number analyzed (Participants) | 55 | 54 | 55 | 55
units on a scale per period | 3.85 (1.95) | 3.58 (1.98) | 3.49 (2.07) | 3.44 (2.00)

6. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Stress.
Description: Stress will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their stress on a scale of 0(low) to 10(high). Levels of EMA stress will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA stress over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA stress will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale per period
Arm/Group | Baseline Assessment Period | Melatonin 3 mg | Melatonin 0.5 mg | Placebo Pill
Number analyzed (Participants) | 55 | 54 | 55 | 55
units on a scale per period | 3.19 (1.86) | 3.34 (1.78) | 3.29 (1.86) | 3.33 (1.96)

7. Secondary Outcome: Mean Fitbit Device Adherence Rate.
Description: For each participant, the proportion of days where the Fitbit device was worn will be calculated. Proportion of days where the Fitbit device was worn across all participants will be reported with means and standard deviations.
Time Frame: as for outcome 1
Population: Pre-specified to report results at the whole sample level. Of the 60 enrolled participants, 55 (91.7%) had sufficient Fitbit data across the 98 day study to include in analyses.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 55
days | 88.01 (3.00)

8. Secondary Outcome: Mean Participant Adherence to Nightly Melatonin 0.5 mg Supplement.
Description: For each participant, the proportion of days where the melatonin 0.5 mg supplement was administered will be calculated. Proportion of days adherent across all participants will be reported with means and standard deviations.
Time Frame: Assessed across the two 14-day treatment periods (28 days total).
Population: Pre-specified to report results at the whole sample level. Of the 60 enrolled participants, 55 (91.7%) had sufficient supplement adherence data across each 28 day study period (3 mg melatonin, .5 mg melatonin, and placebo) to include in analyses.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 55
days | 21.82 (2.19)

9. Secondary Outcome: Mean Participant Adherence to Nightly Melatonin 3 mg Supplement.
Description: For each participant, the proportion of days where the melatonin 3 mg supplement was administered will be calculated. Proportion of days adherent across all participants will be reported with means and standard deviations.
Time Frame: Assessed across the two 14-day treatment periods (28 days total).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 55
days | 21.78 (2.20)

10. Secondary Outcome: Mean Participant Adherence to Nightly Placebo Supplement.
Description: For each participant, the proportion of days where the placebo supplement was administered will be calculated. Proportion of days adherent across all participants will be reported with means and standard deviations.
Time Frame: Assessed across the two 14-day treatment periods (28 days total).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 55
days | 21.53 (2.23)

11. Other Pre Specified Outcome: Mean Within-Subject Difference in Self-Reported Sleep Disturbance.
Description: Participants will rate their sleep disturbance using the Insomnia Severity Index (ISI) administered daily during baseline and intervention periods (14 weeks). Items are rated from 0 to 4, with higher scores indicating greater levels of sleep disturbance. Levels of daily sleep disturbance will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in sleep disturbance over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Difference in self-reported sleep disturbance will be assessed every two weeks between baseline and intervention periods (14 weeks total).
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Within-Subject Difference in Self-Reported Side Effects.
Description: Participant self-reported side effects will be assessed utilizing a weekly survey measure. Number of side effects will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate a count of self-reported side effects in each study period. Side effects over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Self-reported side effects will be assessed via weekly survey during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Pain.
Description: . Pain will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their pain on a scale of 0(low) to 10(high). Levels of EMA pain will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA pain over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA pain will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Mood.
Description: Mood will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0(poor) to 10(excellent). Levels of EMA mood will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA mood over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA mood will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Concentration.
Description: Concentration will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0(low) to 10(high). Levels of EMA concentration will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA concentration over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA concentration will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Confidence.
Description: Confidence will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0(low) to 10(high). Levels of EMA confidence will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Changes in EMA confidence over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA confidence will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Within-Subject Difference in Fitbit Device-Recorded Daily Steps.
Description: . Daily step counts will be assessed by a Fitbit device. Daily step counts will be aggregated within the baseline assessment period and in each of the intervention periods (3 mg melatonin, 0.5 mg melatonin, placebo) to generate an overall mean and standard deviation for each period. Daily steps values over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Daily steps will be assessed consistently via Fitbit device during the baseline assessment period (2 weeks) and during each of the 6 intervention periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Mean Participant Survey Adherence Rate.
Description: For each participant of the proportion of surveys measures completed (both daily and weekly surveys) will be calculated. Proportion of days adherent across all participants will be reported with means and standard deviations.
Time Frame: as for outcome 1
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Mean Participant Ecological Momentary Assessment (EMA) Adherence Rate.
Description: For each participant of the proportion of EMA measures completed will be calculated. Proportion of days adherent across all participants will be reported with means and standard deviations.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data for each participant were collected over a 14-week period (2-week baseline and 12-week intervention).
Description: Systematic assessment was conducted via a daily survey sent to participants asking if they are experiencing any side effects.
Groups:
- 3 mg Melatonin: Dietary Supplement: Melatonin 3 mg
  Participants provided with a smart pill bottle containing a 4-week supply of 3 mg melatonin pills.
- .5 mg Melatonin: Dietary Supplement: Melatonin 0.5 mg
  Participants provided with a smart pill bottle containing a 4-week supply of 0.5 mg melatonin pills.
- Placebo: Cellulose placebo pill
  Participants provided with a smart pill bottle containing a 4-week supply of cellulose placebo pills.
Arm/Group | 3 mg Melatonin | .5 mg Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 3/60 | 0/60 | 0/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg Melatonin (N=60) | .5 mg Melatonin (N=60) | Placebo (N=60)
Headache (General disorders) | 3 (8) | 0 (0) | 0 (0) — Systematic assessment conducted via a daily survey sent to participants asking if they are experiencing any side effects believed to be related to their study pill.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT05349188/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT05349188/ICF_001.pdf